CLINICAL TRIAL: NCT00492323
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group With a Crossover Confirmation Period Study of RWJ-333369 for the Treatment of Postherpetic Neuralgia.
Brief Title: An Effectiveness and Safety Study With RWJ-333369 (Carisbamate) for the Study of Postherpetic Neuralgia (PHN).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR010363; 333369NPP2001
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Postherpetic Neuralgia; Neuralgia; Herpes Zoster
Keywords: pain following the healing of rashes and blisters; herpes virus; rash; varicella-zoster virus; shingles.
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia; Herpes Zoster; Blister; Exanthema; Chickenpox | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 002 (Placebo Comparator): placebo twice daily for 4 weeks
  Interventions: Drug: placebo
- 001 (Experimental): carisbamate 200 mg tablet twice daily for 4 weeks
  Interventions: Drug: carisbamate

INTERVENTIONS:
Drug: placebo — twice daily for 4 weeks
  Arms: 002
Drug: carisbamate — 200 mg tablet twice daily for 4 weeks
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness, and tolerability of 200 mg of RWJ-333369 given twice daily compared with placebo in the treatment of postherpetic neuralgia.

DETAILED DESCRIPTION:
Postherpetic neuralgia is a distressing syndrome of neuropathic pain that continues for at least 3 months after the resolution of the varicella-zoster rash (shingles), can last up to years later, and for which therapies are often limited by incomplete pain relief and side effects. This is a randomized (study medication is assigned by chance), double-blind (neither the Investigator or the patient know the name of the assigned study medication), placebo-controlled, crossover, parallel-group, multicenter study to determine the effectiveness and safety of 200 mg of RWJ-333369 given twice daily for 4 weeks compared with placebo in patients with Postherpetic Neuralgia (PHN). The study hypothesis is that 200 mg of RWJ-333369 given twice daily for 4 weeks will be more effective than placebo in reducing pain due to PHN, as measured by average daily PHN pain scores. Patients will receive 200 mg of RWJ-333369 or matching placebo tablets, given in equally divided doses twice daily by mouth, with or without food, for 4 weeks in each of the 2 treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of postherpetic neuralgia (PHN) with a history of varicella-zoster rash (shingles), persistent pain for at least 6 months after the healing of the rash
* Experienced postherpetic neuralgia pain on a daily basis for the past 3 months
* Women must be postmenopausal for at least 2 years, sexually abstinent, or if sexually active, be practicing an effective method of birth control, and have a negative serum pregnancy test at screening.

Exclusion Criteria:

* History of a poor response to 3 or more medications for postherpetic neuralgia (PHN), with poor response defined as treatment with medications in the following categories of therapy for at least 1 month at therapeutic dosages without at least moderate improvement, as judged by the study doctor: Antiepileptic drugs, antidepressants, serotonin norepinephrine uptake inhibitors (SNRIs), opioid analgesics, or lidocaine patch
* currently taking tricyclic antidepressants, Coumadin (warfarin), or continued treatment with an antiepileptic drug for any indication, Note: If taking these medications, to be eligible for the study, they must be tapered and discontinued
* past neurolytic treatment (destruction of nerves by the application of chemicals, heat or cold, neurosurgery, intrathecal pumps, or spinal cord stimulators for PHN pain
* currently using herbal topical creams or ointments for pain relief within 48 hours, capsaicin within 6 months, or systemic corticosteroids within 3 months of the baseline period
* Prior exposure to RWJ-333369 (carisbamate).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The mean of the last 7 average daily PHN scores of the first treatment period on days when study drug is taken. | 4 weeks

SECONDARY OUTCOMES:
The means of the last 7 average daily PHN pain scores with no use of rescue medication, the last 7 current daily PHN pain scores, the last 7 maximum daily PHN pain scores and the last 7 daily sleep interference scores. | 4 weeks (2 four-week treatment periods (cross-over design )

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.